CLINICAL TRIAL: NCT06178393
Title: Real-World Use of Novel Treatments in Patients With Spinal Muscular Atrophy (SMA): A Multi-Site Retrospective Chart Review of Pediatric SMA Patients Outside of the United States
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COAV101A12402
Record Dates: First submitted 2023-12-11; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (6):
- OA monotherapy
- Nusinersen monotherapy
- Other DMTs switched to OA
- OA add-on other DMTs
- Combination, other DMTs with OA
- Other treatment sequence

SUMMARY:
This global, retrospective, non-interventional, medical chart review (MCR), descriptive study collected patient-level data in regions outside the US.

The study required a repeated data collection at follow-up dates from start of treatment with nusinersen, onasemnogene abeparvovec-xioi (OA), and/or risdiplam. At the start of data collection, the study team reached out to the health care providers (HCPs) involved in treating pediatric SMA patients for participating in this study. The physicians across the participating countries conducted a retrospective MCR of pediatric patients diagnosed with SMA who were treated with at least 1of the 3 novel disease-modifying treatments (DMTs): nusinersen, OA, and/or risdiplam.

All health care encounters data i.e., emergency and inpatient admissions, surgery, and outpatient consultations of recruited patients, including their treatment with nusinersen, OA, and/or risdiplam, were abstracted to understand the treatment patterns as per routine clinical practice for SMA management globally. The first date of initial administration of 1 of the 3 target drugs was used as the "index date." Based on this, the record abstraction was performed through a retrospective MCR during the pre-index period, at index date and in the post-index period.

ELIGIBILITY:
Inclusion criteria:

* Genetically confirmed diagnosis of SMA.
* Aged less than 5 years at index date.
* Initiated treatment with nusinersen or onasemnogene abeparvovec-xioi or risdiplam or any combination of them during the identification period.
* Availability of medical information in chart for at least 1 visit prior to initiation of treatment with the target treatment(s).

Exclusion criteria:

None

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Number and proportion of male patients | Baseline
Number and proportion of female patients | Baseline
Number and proportion of patients per race | Baseline
Number and proportion of patients per insurance type | Baseline
Number and proportion of patients per gestational age category at birth | Baseline
Number and proportion of patients per country | Baseline
Number and proportion of patients with prenatal screening performed and confirmed for SMA | Baseline
Number and proportion of patients undergoing newborn screening for SMA | Baseline
Number and proportion of patients experiencing SMA-related symptoms prior to initiation of the first DMT (index drug) | Baseline
Mean age at onset of SMA-related symptoms experienced prior to initiation of the first DMT | Baseline
Mean age at SMA genetic diagnosis | Baseline
Number and proportion of patients who had as survival of motor neuron 1 (SMN1) genetic test | Baseline
Number and proportion of patients per SMN1 genetic test result category | Baseline
Number and proportion of patients who had a survival of motor neuron 2 (SMN2) genetic test | Baseline
Number and proportion of patients per SMN2 gene copy number | Baseline
Number and proportion of patients per SMA type at diagnosis | Baseline
Mean body weight | Baseline

SECONDARY OUTCOMES:
Time to first improvement from last pre-index/pre-switch assessment | Up to approximately 5 years
Time from pre-index/last pre- switch until the last follow-up visit with available data for the overall developmental motor milestones rates | Up to approximately 5 years
Number and proportion of patients who achieved at least once ≥ 1 point increase on the Hammersmith infant neurological examination: Section 2 (HINE-2, motor milestones) | Up to approximately 5 years
  The HINE-2 assesses motor milestones and includes 8 categories: voluntary grasp, ability to kick in supine position, head control, rolling, sitting, crawling, standing, and walking. Overall scores can range from 0 to 26. Higher scores indicate higher levels of motor ability.
Number and proportion of patients who achieved at least once ≥ 3 points increase on the Hammersmith Functional Motor Scale-Expanded (HFMSE) | Up to approximately 5 years
  The HFMSE is a validated SMA specific assessment devised for use in children with SMA to give objective information on motor ability and clinical progression. The HFMSE contains 33 items rated from 0 (unable to perform) to 2 (performs without modification/adaptation/compensation). Total scores range from 0-66. Higher scores indicate higher levels of motor ability.
Number and proportion of patients who achieved at least once ≥ 3 points decrease on the HFMSE | Up to approximately 5 years
  The HFMSE is a validated SMA specific assessment devised for use in children with SMA to give objective information on motor ability and clinical progression. The HFMSE contains 33 items rated from 0 (unable to perform) to 2 (performs without modification/adaptation/compensation). Total scores range from 0-66. Higher scores indicate higher levels of motor ability.
Number and proportion of patients who maintained score change ±3 points on the HFMSE | Up to approximately 5 years
  The HFMSE is a validated SMA specific assessment devised for use in children with SMA to give objective information on motor ability and clinical progression. The HFMSE contains 33 items rated from 0 (unable to perform) to 2 (performs without modification/adaptation/compensation). Total scores range from 0-66. Higher scores indicate higher levels of motor ability.
Change in score per month on the HFMSE | Baseline up to approximately 5 years
  The HFMSE is a validated SMA specific assessment devised for use in children with SMA to give objective information on motor ability and clinical progression. The HFMSE contains 33 items rated from 0 (unable to perform) to 2 (performs without modification/adaptation/compensation). Total scores range from 0-66. Higher scores indicate higher levels of motor ability.
Estimate of HFMSE score per timepoint during the post period, adjusted for the last pre-value | Up to approximately 15 years
  The HFMSE is a validated SMA specific assessment devised for use in children with SMA to give objective information on motor ability and clinical progression. The HFMSE contains 33 items rated from 0 (unable to perform) to 2 (performs without modification/adaptation/compensation). Total scores range from 0-66. Higher scores indicate higher levels of motor ability.
Number and proportion of patients who achieved at least once ≥ 1 point increase on the Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND) | Up to approximately 5 years
  CHOP INTEND scores can range from 0 to 64, where 64 is the maximum possible score. A higher score indicates higher/better motor function.
Number and proportion of patients who achieved at least once ≥4 points increase on the CHOP INTEND | Up to approximately 5 years
  CHOP INTEND scores can range from 0 to 64, where 64 is the maximum possible score. A higher score indicates higher/better motor function.
Change in score per month on the CHOP INTEND | Baseline up to approximately 5 years
  CHOP INTEND scores can range from 0 to 64, where 64 is the maximum possible score. A higher score indicates higher/better motor function.
Estimate of score per timepoint during the post period, adjusted for the last pre-value on the CHOP INTEND | Up to approximately 15 years
  CHOP INTEND scores can range from 0 to 64, where 64 is the maximum possible score. A higher score indicates higher/better motor function.
Number and proportion of patients without any craniofacial deficits during the post-index period | Up to approximately 15 years
Number and proportion of patients who exhibited at least 1 craniofacial deficit during the post-index period including reduced mouth opening, overbite, narrow/high arched palate, and other craniofacial deficits | Up to approximately 15 years
Number and proportion of patients who remained free of any non-oral support during the post-index period | Up to approximately 15 years
Number and proportion of patients who did not remain free of any non-oral support during the post-index period | Up to approximately 15 years
Number and proportion of patients who exhibited constipation at least once during the post-index period | Up to approximately 15 years
Number and proportion of patients who exhibited failure to thrive or underweight at least once during the post-index period | Up to approximately 15 years
Number and proportion of patients per the Pediatric-Functional Oral Intake Scale (p-FOIS) score at the timepoints of interest | Baseline, 3, 6, and 12 months
  The p-FOIS score has a range of 1 (nothing taken orally) to 6 (age-appropriate oral intake).
Number and proportion of patients who had improvement (the p-FOIS score increased by at least 1 point between the timepoints of interest) | Baseline, 3, 6, and 12 months
  The p-FOIS score has a range of 1 (nothing taken orally) to 6 (age-appropriate oral intake).
Number and proportion of patients who had decline (the p-FOIS score decreased by at least 1 point between the timepoints of interest) | Baseline, 3, 6, and 12 months
  The p-FOIS score has a range of 1 (nothing taken orally) to 6 (age-appropriate oral intake).
Number and proportion of patients who maintained status (the p-FOIS score maintained stable between the timepoints of interest) | Baseline, 3, 6, and 12 months
  The p-FOIS score has a range of 1 (nothing taken orally) to 6 (age-appropriate oral intake).
Number and proportion of patients with unknown status (unknown/missing p-FOIS score in any of the timepoints of interest) | Baseline, 3, 6, and 12 months
  The p-FOIS score has a range of 1 (nothing taken orally) to 6 (age-appropriate oral intake).
Number and proportion of patients with p-FOIS <3 at the timepoints of interest in the functional swallow category | Baseline, 3, 6, and 12 months
  The p-FOIS score has a range of 1 (nothing taken orally) to 6 (age-appropriate oral intake).
Number and proportion of patients with p-FOIS ≥ 3 at the timepoints of interest in the functional swallow category | Baseline, 3, 6, and 12 months
  The p-FOIS score has a range of 1 (nothing taken orally) to 6 (age-appropriate oral intake).
Number and proportion of patients who achieved (patients who went from the p-FOIS < 3 to the p-FOIS ≥ 3 category between the timepoints of interest) in the functional swallow category | Baseline, 3, 6, and 12 months
  The p-FOIS score has a range of 1 (nothing taken orally) to 6 (age-appropriate oral intake).
Number and proportion of patients who lost (patients who went from the p-FOIS ≥ 3 to p-FOIS <3 category between the timepoints of interest) in the functional swallow category | Baseline, 3, 6, and 12 months
  The p-FOIS score has a range of 1 (nothing taken orally) to 6 (age-appropriate oral intake).
Number and proportion of patients who maintained status (patients who remained at p-FOIS <3 category between the timepoints of interest) in the functional swallow category | Baseline, 3, 6, and 12 months
  The p-FOIS score has a range of 1 (nothing taken orally) to 6 (age-appropriate oral intake).
Number and proportion of patients who maintained status (patients who remained at p-FOIS ≥ 3 category between the timepoints of interest) in the functional swallow category | Baseline, 3, 6, and 12 months
  The p-FOIS score has a range of 1 (nothing taken orally) to 6 (age-appropriate oral intake).
Number and proportion of patients with unknown (unknown/missing p-FOIS score in any of the timepoints of interest) in the functional swallow category | Baseline, 3, 6, and 12 months
  The p-FOIS score has a range of 1 (nothing taken orally) to 6 (age-appropriate oral intake).
Number and proportion of patients with p-FOIS <4 at the timepoints of interest in the total oral nutrition category | Baseline, 3, 6, and 12 months
  The p-FOIS score has a range of 1 (nothing taken orally) to 6 (age-appropriate oral intake).
Number and proportion of patients with p-FOIS ≥ 4 at the timepoints of interest in the total oral nutrition category | Baseline, 3, 6, and 12 months
  The p-FOIS score has a range of 1 (nothing taken orally) to 6 (age-appropriate oral intake).
Number and proportion of patients who achieved (patients who went from the p-FOIS <4 to p-FOIS ≥ 4 category between the timepoints of interest) in the total oral nutrition category | Baseline, 3, 6, and 12 months
  The p-FOIS score has a range of 1 (nothing taken orally) to 6 (age-appropriate oral intake).
Number and proportion of patients who lost (patients who went from the p-FOIS ≥ 4 to p-FOIS <4 category between the timepoints of interest) in the total oral nutrition category | Baseline, 3, 6, and 12 months
  The p-FOIS score has a range of 1 (nothing taken orally) to 6 (age-appropriate oral intake).
Number and proportion of patients who maintained status (patients who remained at p-FOIS< 4 category between the timepoints of interest) in the total oral nutrition category | Baseline, 3, 6, and 12 months
  The p-FOIS score has a range of 1 (nothing taken orally) to 6 (age-appropriate oral intake).
Number and proportion of patients who maintained status (patients who remained at p-FOIS≥ 4 category between the timepoints of interest) in the total oral nutrition category | Baseline, 3, 6, and 12 months
  The p-FOIS score has a range of 1 (nothing taken orally) to 6 (age-appropriate oral intake).
Number and proportion of patients with unknown status (unknown/missing p-FOIS score in any of the timepoints of interest) in the total oral nutrition category | Baseline, 3, 6, and 12 months
  The p-FOIS score has a range of 1 (nothing taken orally) to 6 (age-appropriate oral intake).
Number and proportion of patients without any swallow evaluation during the post-index period | Up to approximately 15 years
Number and proportion of patients with at least 1 swallow evaluation during the post index period including the type of swallow evaluation | Up to approximately 15 years
Number and proportion of patients with at least 1 symptom of interest related to eating during the post-index period | Up to approximately 15 years
  Symptoms of interest were coughing/choking with liquids; coughing/choking with solids; prolonged feeding times; fatigue with eating; swallowing or feeding difficulties; difficulty chewing; and wet/gurgles after eating.
Number and proportion of patients without any sign of aspiration during the post-index period | Up to approximately 15 years
Number and proportion of patients with at least 1 aspiration sign during the post-index period for each of the following consistencies: thin liquids; nectar liquids (mildly thick); honey liquids (moderately thick); puree; solid | Up to approximately 15 years
Number and proportion of patients without any deficits in swallowing during the post-index period | Up to approximately 15 years
Number and proportion of patients who exhibited nasal regurgitation at least once during the post-index period | Up to approximately 15 years
Number and proportion of patients who exhibited no swallow initiation at least once during the post-index period | Up to approximately 15 years
Number and proportion of patients who exhibited pharyngeal residue at least once during the post-index period | Up to approximately 15 years
Number and proportion of patients who exhibited aspiration at least once during the post-index period | Up to approximately 15 years
Number and proportion of patients who suffered penetration at least once during the post-index period | Up to approximately 15 years
Number and proportion of patients who were able to drink thin liquids during the post-index period | Up to approximately 15 years
Number and proportion of patients who were able to drink thin nectar during the post-index period | Up to approximately 15 years
Number and proportion of patients who were able to drink nectar during the post-index period | Up to approximately 15 years
Number and proportion of patients who were able to drink honey during the post-index period | Up to approximately 15 years
Number and proportion of patients who reported at least once the following deficits relating to the patients cry/voice during the post-index period: not audible; quiet/weak/hard to hear; wet/gurgly; breathy; unknown/not reported | Up to approximately 15 years
Number and proportion of patients who did not experience fatigue with speech over the course of the day during the post-index period | Up to approximately 15 years
Number and proportion of patients who experienced at least once fatigue with speech over the course of the day during the post-index period | Up to approximately 15 years
Number and proportion of patients who experienced at least once clinical signs of aspiration during the post-index period | Up to approximately 15 years
Number and proportion of patients who experienced at least once problem in chewing during the post-index period | Up to approximately 15 years
Number and proportion of patients who experienced at least once aversion/disinterest in eating or drinking | Up to approximately 15 years
Number and proportion of patients who experienced at least once a concern for insufficient oral nutrient ingestion | Up to approximately 15 years
Number and proportion of patients per category of maximum speech milestone achieved during the post-index period. | Up to approximately 15 years
Number and proportion of patients who experienced clinical signs of aspiration at the timepoints of interest | Baseline, 3, 6, and 12 months
Number and proportion of patients with improvement (patients who had clinical signs of aspiration at the first timepoint of interest and lost it at the next timepoint of interest) | Baseline, 3, 6, and 12 months
Number and proportion of patients with decline (patients who didn't have any clinical signs of aspiration at the first timepoint of interest and gained it at the next timepoint of interest) | Baseline, 3, 6, and 12 months
Number and proportion of patients who maintained status (patients without clinical signs of aspiration at both timepoints of interest) | Baseline, 3, 6, and 12 months
Number and proportion of patients who maintained status (patients with clinical signs of aspiration at both timepoints of interest) | Baseline, 3, 6, and 12 months
Number and proportion of patients with unknown status (patients with unknown/missing clinical signs of aspiration in any of the timepoints of interest) | Baseline, 3, 6, and 12 months
Number and proportion of patients who experienced fatigue with eating at the timepoints of interest | Baseline, 3, 6, and 12 months
Number and proportion of patients with improvement (patients who experienced fatigue with eating at the first timepoint of interest and did not experience it at the next timepoint of interest) | Baseline, 3, 6, and 12 months
Number and proportion of patients with decline (patients who didn't experience fatigue with eating at the first timepoint of interest and experienced it at the next timepoint of interest) | Baseline, 3, 6, and 12 months
Number and proportion of patients who maintained status (patients who didn't experience fatigue with eating at both timepoints of interest) | Baseline, 3, 6, and 12 months
Number and proportion of patients who maintained status (patients who experienced fatigue with eating at both timepoints of interest) | Baseline, 3, 6, and 12 months
Number and proportion of patients with unknown status (patients with unknown/missing experience of fatigue with eating in any of the timepoints of interest) | Baseline, 3, 6, and 12 months
Number and proportion of patients per each category of maximum speech milestone achieved at the timepoints of interest | Baseline, 3, 6, and 12 months
Number and proportion of patients with improvement (patients who had cooing as a maximum speech milestone at the first timepoint of interest and achieved at least 1 more speech milestone at the next timepoint of interest) | Baseline, 3, 6, and 12 months
Number and proportion of patients with decline in speech milestones | Baseline, 3, 6, and 12 months
  Decline was defined as patients who had consonant and vowel combination; babbling word(s); combining 2 words together; speech understood by family members; or speech understood by unfamiliar listeners as a maximum speech milestone at the first timepoint of interest and cooing at the next timepoint of interest.
Number and proportion of patients who maintained status (patients who remained at cooing between the timepoints of interest or patients who remained at 'consonant and vowel combination' or above between the timepoints of interest) | Baseline, 3, 6, and 12 months
Number and proportion of patients with unknown status (patients with unknown/missing maximum speech milestone in any of the timepoints of interest) | Baseline, 3, 6, and 12 months
Number and proportion of patients with normal pulmonary evaluation during the post-index period | Up to approximately 15 years
Number and proportion of patients with at least 1 abnormal pulmonary evaluation during the post-index period | Up to approximately 15 years
Number and proportion of patients who experienced at least once chest abnormality symptoms during the post-index period | Up to approximately 15 years
Number and proportion of patients who experienced at least once pneumonia or respiratory illness during the post-index period | Up to approximately 15 years
Number and proportion of patients who experienced at least once paradoxical breathing symptoms during the post-index period | Up to approximately 15 years
Number and proportion of patients who used sitting and mobility support devices during the post-index period | Up to approximately 15 years
Number and proportion of patients who used at least once the following sitting and mobility support devices during the post-index period: standing frame; positioning device; adaptive seating system; gait trainer; walker; wheelchair; scooter; other | Up to approximately 15 years
Time from index date to the first initial improvement in motor function | Up to approximately 15 years
Number and proportion of patients who had overall improvement at the end of post-index period as per physicians' assessment for general impression, motor function, respiratory function, and swallow function | Up to approximately 15 years
Number and proportion of patients per survival status | Up to approximately 15 years
Number and proportion of patients per cause of death | Up to approximately 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, Bannockburn, Illinois, United States